CLINICAL TRIAL: NCT06361654
Title: Effect of Muscular Imbalance Between Flexors and Extensors of the Fingers and Wrist on Upper Limb Injuries in Climbers, a Longitudinal Study.
Brief Title: Effect of Muscular Imbalance Between Flexors and Extensors of the Fingers and Wrist on Upper Limb Injuries in Climbers
Acronym: CRIMPER
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/0135/OB
Record Dates: First submitted 2024-03-22; First posted 2024-04-12 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-03

CONDITIONS: Climber

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: The strength values of the flexors and extensors of the fingers and wrist will be measured using a dynamometer — The measurements will be taken during different climbing sessions, after the warm-up.
  The study will include measurements on different climbers. Informed consent and personal data will be collected from the climbers before the measurements are taken. The strength values of the flexors and extensors of the fingers and wrist will be measured using a dynamometer.

SUMMARY:
Climbing is a booming sport with an increasing number of participants. When practicing this sport, there is a muscular imbalance between the flexor and extensor systems (especially in the fingers), with the flexors of the fingers exerting greater force than the extensors. In addition, upper limb injuries, particularly the fingers, are very common.

The study will be carried out on club-licensed climbers, as they are better supervised. They will be recruited through requests sent to various clubs. The measurements will be taken during different climbing sessions, after the warm-up.

The study will include measurements on different climbers. Informed consent and personal data will be collected from the climbers before the measurements are taken. The strength values of the flexors and extensors of the fingers and wrist will be measured using a dynamometer. The climbers will then continue their usual training for 1 year. For 1 year after the measurements, the climbers will be contacted every month by telephone to collect the different injuries they may have suffered in relation to climbing, as well as the number of hours they have spent climbing in the past month. After 1 year, the annual number of hours of climbing and the annual number of injuries can be calculated for each climber. Injury is defined as any medically diagnosed lesion of the musculoskeletal system of the upper limb or pain that prevents the practice of a sport whose aetiology is climbing. These data are used to calculate the "athlete exposure" (A-E), i.e. the incidence of injury per 1000 hours of practice. As the study population is large, this allows for variations in exposure between subjects.

ELIGIBILITY:
* A male or female climber who has been a member of a climbing club for at least 1 year;
* Have a level of 6a "on sight" or higher;
* Fluent in spoken and written French;
* Over 18 years of age.

Exclusion Criteria:

* Declaration of a medically diagnosed upper limb injury at the time of testing;
* Presence of any pathology that prevents climbing or taking finger or wrist measurements;
* Volunteers for whom it is impossible to collect data by telephone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: climber
Sampling Method: Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-03-25 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Athlete exposure | through study completion, an average of 1 year
  - Athlete exposure (A-E): the incidence of climbing-related upper limb injuries reported over 1000 climbing hours (declarative). The number of injuries and climbing hours will be collected by telephone every month for 1 year;

CONTACTS AND LOCATIONS:
Locations (1):
- Rouen, University Hospital, Rouen, Normandy, France

IPD SHARING:
Plan to Share IPD: No